CLINICAL TRIAL: NCT02146391
Title: AN OPEN-LABEL, RANDOMIZED, SINGLE-DOSE, TWO-WAY CROSSOVER STUDY TO EVALUATE THE EFFECT OF FOOD UPON THE PHARMACOKINETICS OF ANDROXAL
Brief Title: Study to Evaluate the Effect of Food Upon the Pharmacokinetics of Androxal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZA-107
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Normal Volunteers
MeSH Terms: interventions — Enclomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Androxal 25 mg (Experimental)
  Interventions: Drug: Androxal 25 mg Capsules

INTERVENTIONS:
Drug: Androxal 25 mg Capsules

SUMMARY:
This study is an open-label, randomized, single-center, single-dose, two-way crossover study of the PK properties of Androxal in healthy male subjects. Twelve male subjects will each receive a single dose of Androxal 25 mg in both the fed and fasting state.

ELIGIBILITY:
Inclusion Criteria:

1. Speak, read, and understand English or Spanish and is willing and able to provide written informed consent on an IRB-approved form prior to the initiation of any study procedures;
2. Male; age 18-60 with a BMI of 25-42 kg/m2 inclusive
3. No significant abnormal findings at the screening physical examination as evaluated by the Investigator;
4. Normal laboratory values (or abnormal but not clinically significant) at screening as determined by the Investigator;
5. Subject is willing to remain in the clinic for the screening visit and 2 overnight treatment visits (approximately 36 hours for the treatment visit)
6. Must be able to swallow gelatin capsules;
7. Must be willing to remain in the clinic for the treatment visits

Exclusion Criteria:

1. Known hypersensitivity to Clomid;
2. Abnormal screening visit vital signs or clinical laboratory evaluation considered clinically significant by the Investigator;
3. A hematocrit >54% or a hemoglobin >17 g/dL.
4. Subject with a significant organ abnormality or disease as determined by the Investigator;
5. Any medical condition that would interfere with the study as determined by the Investigator;
6. Participation in a clinical trial with investigational medication within 30 days prior to study medication administration;
7. An acute illness within 5 days of study medication administration;
8. Positive urine drug screen at the screening visit;
9. Known history of HIV and/or Hepatitis B or C
10. Tobacco (nicotine products) use in the 3 months prior to the study;
11. A mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study and/or evidence of an uncooperative attitude, as determined by the Investigator;
12. History of venous thromboembolic disease (e.g. deep vein thrombosis or pulmonary embolism);
13. History of myocardial infarction, unstable angina, symptomatic heart failure, ventricular dysrhythmia, or known history of QTc interval prolongation;
14. An employee or family member of an employee of the study site or the Sponsor;
15. Previous participation in a clinical study of Androxal.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
• Cmax of a single dose of 25 mg of Androxal in male subjects in the fed state and fasted state. | 24 hour